CLINICAL TRIAL: NCT04136015
Title: A Prospective Study on Early Conversion of Dasatinib in CML-CP Patients Who Have Not Early Molecular Response on Imatinib
Brief Title: Early Conversion of Dasatinib in CML-CP Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, xuna, Associate chief physician, Nanfang Hospital, Southern Medical University
Other Study IDs: TKIs-cml-001
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Validity and Safety
MeSH Terms: interventions — Dasatinib

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dasatinib group
  Interventions: Drug: Dasatinib 100 MG
- Imatinib group
  Interventions: Drug: Dasatinib 100 MG

INTERVENTIONS:
Drug: Dasatinib 100 MG — The CML-CP patients with early(3m to 6m) molecular response failure on imatinib,Conversion dasatinib group or Imatinib group

SUMMARY:
Chronic myeloid leukemia (CML) is a malignant disease of acquired hematopoietic stem cells. The BCR-ABL fusion gene is the pathogenic basis of CML. Tyrosine kinase inhibitors (TKIs) are targeted drugs for this fusion protein. With the wide clinical application of TKIs, the efficacy of CML patients has been greatly improved. However, there are still a significant number of patients who have poor response to the first generation of TKI drugs, imatinib, most of them have early molecular response failures (BCR-ABL（IS）>10% at 3 or 6 months) ，which means lower rates of molecular response, increased risk of progression, and higher overall survival. For them, the early conversion of dasatinib might be a better choice.

ELIGIBILITY:
Inclusion Criteria:

1.18-65 years old； 2.CML-CP,and Imatinib treatment longest for 6 months ； 3.Q-pcr monitoring of BCR/ABLIS failed to achieve the best therapeutic effect（BCR/ABLIS>10.00% in 3m or BCR/ABLIS>1.00% in 6m）； 4.No previous history of malignant tumor; 5.Informed consent of the patient or his legal representative

Exclusion Criteria:

1. History of CML-CP or CML-AP;
2. Resistant to dasatinib,or treatment with imatinib more than 6 months;
3. Received allogeneic hematopoietic stem cell transplantation,or immunotherapy;
4. woman who is pregnant or nursing
5. Combined with other serious organic diseases, serious arrhythmia, pulmonary hypertension, cardiomyopathy, serious autoimmune diseases.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: CML-CP patients treated with imatinib failed to achieve the best therapeutic effect（BCR/ABLIS>10.00% in 3m or BCR/ABLIS>1.00% in 6m）convert to dasatinib.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
MMR in 1 year | 1 year
  MMR(BCR/ABL(IS)<0.1%) at 12 months after switching to dasatinib for patients who did not achieve optimal treatment with imatinib for 3 to 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- NanfangH, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes